CLINICAL TRIAL: NCT00780923
Title: A Longitudinal Study of Short-Term Effects of CPAP Treatment on Airway and Systemic Inflammation in Patients With Obstructive Sleep Apnea
Brief Title: Effect of Continuous Positive Airway Pressure Treatment on Inflammation in Patients With Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyoto University, Graduate School of Medicine (Other)
Responsible Party: Principal Investigator, Toru Oga, Associate Professor, Respiratory Care and Sleep Control Medicine, Kyoto University Graduate School of Medicine, Kyoto University, Graduate School of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E-558
Record Dates: First submitted 2008-10-27; First posted 2008-10-28 (Estimated); Last update posted 2013-03-27 (Estimated); Status verified 2013-03

CONDITIONS: Obstructive Sleep Apnea; Inflammation; Continuous Positive Airway Pressure
MeSH Terms: conditions — Sleep Apnea, Obstructive; Inflammation | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CPAP (Experimental)
  Interventions: Device: CPAP treatment

INTERVENTIONS:
Device: CPAP treatment — maintains upper airway patency and minimizes the obstructive events
  Other Names: REMstar(Respironics), SleepMate(ResMed)

SUMMARY:
The purpose of this study is to evaluate the effects of CPAP treatment on airway and systemic inflammation in obstructive sleep apnea.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is characterised by repetitive episodes of upper airway obstruction during sleep. Systemic and airway inflammation has been recently shown to be associated with OSA and is hypothesized to contribute to the clinical manifestation and the complications of OSA patients.

Continuous positive airway pressure (CPAP) is a first-line treatment for OSA and improves diurnal and nocturnal symptoms. However, the effectiveness of CPAP in reversing airway inflammation is less compelling in comparison to systemic inflammation.

This study will assess NO in exhaled breath, inflammatory biomarkers in induced sputum and blood of OSA patients and other clinical measurements before and after 3 months of CPAP treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects on admission for sleep study under the Respiratory Care and Sleep Control Medicine, Kyoto University Hospital.
* Subjects diagnosed with OSA (apnea hypopnea index >=20/hour) by overnight polysomnography.

Exclusion Criteria:

* Known history of respiratory diseases that will affect airway inflammatory markers like asthma, chronic obstructive pulmonary disease and bronchiectasis.
* Treatments with corticosteroids or other immunosuppressive drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2009-01; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Inflammatory biomarkers in induced sputum and blood. Cell counts in induced sputum. | 3 months

SECONDARY OUTCOMES:
NO in exhaled breath | 3 months
Airway resistance | 3 months
PSG measurement(AHI,etc.) | 3 months
Quality of Life | 3 months
Psychological status | 3 months
Sleep quality | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Kazuo Chin, MD,PhD, Principal Investigator — Kyoto University, Graduate School of Medicine; Toru Oga, MD,PhD, Principal Investigator — Kyoto University, Graduate School of Medicine
Locations (1):
- Kyoto University Graduate School of Medicine, Kyoto, Kyoto, Japan